CLINICAL TRIAL: NCT06631105
Title: Capability Assessment for Diet and Activity Model Extended to Include Screening and Knowledge in Diabetic Adults
Brief Title: Capability Assessment for Diet and Activity (CADA) Model for Diabetes
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00006976
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: Diabetes; Hospital Admission; Hospital
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates the capabilities related to diet, physical activity, screening, and knowledge among diabetic adults with or without a history of hospital admissions in Central Florida. The hypothesis is that enhancing these capabilities, based on the Capability Approach framework, can significantly reduce hospital readmissions and improve diabetes management outcomes.

DETAILED DESCRIPTION:
Managing diabetes effectively requires a comprehensive understanding of various capabilities, including diet, physical activity, regular screening, and diabetes-related knowledge. For diabetic adults with a history of hospital admissions, these capabilities are critical in preventing readmissions and improving overall health outcomes.

The objective of this study is to extend the investigation of feasible opportunities for managing diabetes by including measures of screening practices and knowledge alongside diet and physical activity. By employing the Capability Approach, this research aims to provide a comprehensive assessment of how these capabilities interact with individual and environmental factors to affect diabetes management. This approach will enrich existing knowledge by highlighting the interplay between diet, activity, screening, and knowledge, and how these factors collectively impact health outcomes. It will also inform targeted interventions that address both personal and environmental determinants of diabetes management, contributing to more effective public health strategies.

The study uses a survey instrument to collect data from diabetic adults who have experienced hospital admissions in Central Florida and those who don't. The data will be analyzed using Structural Equation Modeling (SEM) to explore the relationships and potential causal pathways between the capabilities assessed (diet, activity, screening, knowledge) and health outcomes. This approach, grounded in the Capability Approach framework, will help identify how each capability contributes to the management of diabetes and highlight areas for targeted interventions.

This study is available in English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18.
* Persons diagnosed with diabetes
* Have an email account with access to a reliable internet connection or smartphone

Exclusion Criteria:

* Minors , ages under 18
* Adults not diagnosed with diabetes
* Adults who are unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must be 18 years of age or older and diagnosed with diabetes to take part in this research study . Participants do not need to have ever been hospitalized to take part in this study. Participants will provide informed consent online and complete the survey online at their convenience. This study is available in English and Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
The assessment of relationships between capabilities and health outcomes using the Structural Equation Modeling (SEM) based on the Capability Approach | 1 year
  The research employs a survey instrument with Likert-scale and open-ended questions, targeting diabetic adults with or without previous hospital admissions in Central Florida. Structural Equation Modeling (SEM) based on the Capability Approach will be used to analyze the data, allowing for the examination of relationships between capabilities (diet, activity, screening, knowledge) and health outcomes. The SEM will help identify the direct and indirect effects of these capabilities on diabetes management, providing insights into potential intervention points for improving health outcomes in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States